CLINICAL TRIAL: NCT03529422
Title: A Phase II Study of Durvalumab (MEDI 4736) With Radiotherapy for the Adjuvant Treatment of Intermediate Risk Head and Neck Squamous Cell Carcinoma
Brief Title: Durvalumab With Radiotherapy for Adjuvant Treatment of Intermediate Risk SCCHN
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC1725
Record Dates: First submitted 2018-05-07; First posted 2018-05-18 (Actual); Results first posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Larynx; Lip; Oral Cancer; Digestive Organs--Diseases
Keywords: Head and Neck; Larynx; Lip; Oral Cancer
MeSH Terms: conditions — Laryngeal Diseases; Lymphoid Interstitial Pneumonia; Mouth Neoplasms | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-label, single-arm (Other): Durvalumab in combination with intensity modulated radiotherapy (IMRT) treatments
  Interventions: Drug: Durvalumab; Radiation: Intensity Modulated Radiotherapy Treatments

INTERVENTIONS:
Drug: Durvalumab — Durvalumab 1500mg IV every 3 weeks for 6 cycles
  Other Names: Imfinzi
Radiation: Intensity Modulated Radiotherapy Treatments — Total dose will be 60 Gray (Gy) at 2Gy per fractions for 30 fractions delivered Monday through Friday for 6 weeks
  Other Names: IMRT

SUMMARY:
The purpose of this study is to investigate other drugs that may be combined with radiation to treat cancer. The study focuses on determining whether a combination of durvalumab with radiation can both improve cure rate and at the same time have less serious side effects. Throughout this document, this investigational drug will be referred to as the "study drug", or named individually (durvalumab). The study drug in this research is referred to as investigational because the U.S. Food and Drug Administration (FDA) has not yet approved itfor the treatment of head and neck cancer. Durvalumab was FDA approved in 2017 for the treatment of certain types of bladder cancer, but has not been approved for use in Head and Neck cancer patients.

Durvalumab is an experimental drug that uses the body's immune system to fight the cancer. This study drug is being used in other ongoing clinical trials for other types of cancers. The doctor feels that a patient may experience fewer side effects using this study drug with radiation rather than using cisplatin. The doctor is also investigating whether using this drug can increase the effectiveness of treatment.

DETAILED DESCRIPTION:
Primary Objective -To estimate median 3-year disease free survival (DFS) in patients with intermediate-risk HNSCC treated with adjuvant durvalumab with radiotherapy.

Secondary Objectives

* To characterize safety by evaluating Grade 3-4 acute toxicities of adjuvant durvalumab with radiotherapy in intermediate-risk HNSCC patients
* To characterize the Grade 3-4 chronic toxicities of adjuvant durvalumab with radiotherapy in intermediate-risk HNSCC patients.
* To characterize any-grade chronic toxicities of adjuvant durvalumab with radiotherapy in intermediate-risk HNSCC patients.
* To estimate median OS in patients with intermediate-risk HNSCC treated with adjuvant durvalumab with radiotherapy.
* To correlate PD-L1 expression with disease free survival

Exploratory Objectives

* To analyze disease free survival by HPV status
* To determine how treatment with adjuvant durvalumab and radiotherapy changes markers of tumor infiltrating lymphocytes (TIL)

Primary Endpoint

-3-year DFS will be estimated via the Kaplan-Meier method. DFS is defined as the time from D1 of treatment to time of disease recurrence or death

Secondary Endpoints

* Grade 3-5 acute toxicity will be evaluated according to guidelines from NCI CTCAE, v5.0 and include toxicity from the first day of treatment with immunotherapy until 30 days after completion of concurrent immunotherapy and radiation. Toxicity will include all toxicity attributed to the total study regimen (inclusive of radiation) not just to durvalumab alone.
* Grade chronic 3-5 toxicity will be evaluated according to guidelines from NCI CTCAE, v5.0 and include toxicity continuing or occurring 30 days after completion of concurrent immunotherapy and radiation, and will be followed for up to 6 months.
* OS will be estimated via the Kaplan-Meier method. OS is defined as the time from D1 of treatment to death from any cause.
* Measure PD-LI expression by immunohistochemistry. Pre-treatment PD-L1 expression will be correlated with disease free survival following treatment of adjuvant durvalumab with radiotherapy.

Exploratory Endpoints

* Measure HPV status. HPV status will be correlated with disease free survival following treatment of adjuvant durvalumab with radiotherapy
* Measure tumor infiltrating lymphocytes (TIL) by flow cytometry at baseline (post-surgical, pre-treatment tissue) and at disease progression (post-treatment tissue). Changes in TIL levels will be compared between these two time points.

Treatment Dosage This Phase II trial will evaluate the combination of durvalumab with radiation therapy as post-operative therapy in intermediate risk patients with HNSCC. All patients will receive durvalumab and radiation therapy during cycles 1-3. Radiation therapy is administered per standard radiation oncology regimens, on a daily basis and/or as scheduled during a Monday-Friday working week. Radiation therapy is given concurrently with durvalumab during Cycles 1-3. Durvalumab treatment (1500 mg Q3W) Cycles 1-3 are 3-weeks long cycles (total of 9 weeks). Radiation therapy will be delivered at a dose of 2 Gy over 30 fractions totalling a final dose of 60 Gy. Radiation treatment will take 6 weeks (Mon-Fri) or 30 days and will occur for 6 of 9 weeks that define Cycles 1-3. However, due to delays or missed appointments, completion of those 30 fractions may take longer than the allotted 6 weeks and this is allowed. Radiation therapy must be scheduled and completed within Cycles 1-3 and should not extend into Cycle 4. Please refer to Section 6.2 for additional details and allowances.

During Cycle 4-6, only durvalumab 1500mg Q4W will be given.

Duration of Follow Up All patients will be followed for up to 5 years, or until death, whichever occurs first after removal from study treatment for determination of study endpoints. Patients removed from study treatment for unacceptable adverse event (AE)s will be followed for resolution or stabilization of the adverse event(s). All patients (including those withdrawn for AEs) should be followed after removal from study treatment as stipulated in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained to participate in the study and HIPAA authorization for release of personal health information. Consent for the use of any residual material from biopsy (archival tissue) and serial blood draws will be required for enrollment.
* Age ≥ 18 years of age on day of signing informed consent
* ECOG Performance Status of 0 or 1 (See Appendix 12.4: ECOG Performance Status)
* Histologically confirmed squamous cell carcinoma of the head and neck, including the following subtypes: oral cavity, oropharynx, hypopharynx, larynx
* Must have undergone gross total resection of the primary tumor with curative intent within the past 8 weeks with surgical pathology demonstrating ≥ 1 of the following criteria for "intermediate" risk of recurrence:

  * perineural invasion
  * lymphovascular invasion
  * single lymph node > 3 cm or at least 2 nodes without evidence of extracapsular extension
  * close margins defined as < 5 mm but not frankly positive (in the case of ambiguous, controversial, or superseded margins, final clinical assessment regarding margin status will prevail)
  * pathologically confirmed T3 or T4 primary tumor
* No prior therapy to primary tumor prior to surgical resection (no induction therapy or recurrent disease).
* Demonstrated adequate organ function as defined in the protocol
* Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 7 days prior to treatment. NOTE: Females are considered of child bearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months. Documentation of postmenopausal status must be provided.
* WOCBP must be willing to abstain from heterosexual activity or to use at least 1 highly effective method of contraception from the time of informed consent until 90 days after durvalumab monotherapy treatment is discontinued (whichever is longer). See section 5.6 of the protocol for additional details on contraception requirements for WOCBP and male participants in this trial.
* Male patients with female partners must have had a prior vasectomy or agree to use an adequate method of contraception (i.e., double barrier method: condom plus spermicidal agent) starting with the first dose of study therapy through 90 days after durvalumab monotherapy is discontinued.
* Subjects must be willing and able to comply with study procedures based on the judgment of the investigator or protocol designee.

Exclusion Criteria:

Subjects meeting any of the following exclusion criteria will not be able to participate in this study:

* Is currently participating in or has participated in a study of an investigational agent or an investigational device within 4 weeks of the first dose of treatment.
* Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.
* Has evidence of metastatic disease at time of diagnosis
* Is receiving concurrent chemotherapy, investigational drug, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
* Treatment with any investigational drug within 28 days or 5 half-lives of Day 1 of treatment on this study, whichever is shortest.
* Has not received any antibiotics <7 days prior to 1st dose of durvalumab. If the patient receives either IV antibiotics or >5 day treatment course (oral or IV), then the 1st durvalumab dose should not be given until 14 days of last antibiotic dose. During eligibility screening, subjects who receive any antibiotics within 30 days prior to the proposed initial infusion of durvalumab should be flagged and reviewed by the site's Principle Investigator to determine if the subject is a good candidate to receive durvalumab.
* Known allergy or hypersensitivity to durvalumab or any of the study drug excipients.
* Prior randomization or treatment in a previous durvalumab clinical study regardless of treatment arm assignment.
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

  * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
  * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
* Has received systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Active infection requiring systemic therapy including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies).

  * Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible.
  * Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Has a known contraindication to radiation therapy, including inherited syndromes associated with hypersensitivity to ionizing radiation such as Ataxia-Telangiectasia and Nijmegen Breakage Syndrome
* Has a history of uncontrolled liver disease (including but not limited to cirrhosis).
* Subjects with baseline weight ≤ 40kg (88 lbs).
* Female patients who are pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study) or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy.
* History of another primary malignancy except for.

  * Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease
* History of leptomeningeal carcinomatosis.
* Has an active autoimmune disease (or inflammatory disorders) requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]).

The following are exceptions to this criterion:

* Subjects with vitiligo or alopecia or resolved childhood asthma/atopy
* Subjects who require intermittent use of bronchodilators or local steroid injections would not be excluded from the study.
* Subjects with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement or with Sjorgen's syndrome will not be excluded from the study
* Any chronic skin condition that does not require systemic therapy
* Subjects without active HNSCC disease in the last 5 years may be included but only after consultation with the study physician
* Subjects with celiac disease controlled by diet alone

  * Has a history of non-infectious pneumonitis that required steroids or evidence of interstitial lung disease or current active, non-infectious pneumonitis.
  * Major surgical procedure (as defined by the Investigator) within 21 days prior to the first dose of investigational product (IP). Note: Local surgery of isolated lesions for palliative intent is acceptable.
  * Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
  * Receipt of live attenuated vaccine within 30 days prior to the first dose of study drug. Note: Patients, if enrolled, should not receive live vaccine whilst receiving study treatment and up to 30 days after the last dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2026-05-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Siddharth Sheth, DO MPH, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (3):
- United States (3):
  - University Of Alabama At Birmingham, Birmingham, Alabama
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Medical University of South Carolina - Hollings Cancer Center, Charleston, South Carolina

REFERENCES:
- See also: UNC Lineberger Comprehensive Cancer Center website — http://unclineberger.org/
- See also: North Carolina Cancer Hospital website — http://unclineberger.org/about/nccancerhospital
- See also: National Cancer Institute website — http://www.cancer.gov

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in the study between 10/07/2019 and 05/04/2021 at three cancer centers in the United States.
Period: Overall Study
Arm/Group | Open-label, Single-arm
Started | 18
Completed | 14
Not Completed | 4
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 1
Not completed — Disease progression | 2

BASELINE CHARACTERISTICS:
Arm/Group | Open-label, Single-arm
Number analyzed (Participants) | 18
Age, Continuous [Median (Full Range); unit: years] | 61 [30 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival Rate
Description: Disease-free Survival Rate (DFS) defined as the percentage of participants who were disease-free and alive at 3 years, counting the time from day 1 of treatment to time of disease recurrence or death, was calculated based on the Kaplan-Meier method.
Time Frame: 3 years
Population: Participants started to study treatment and treatment responses were assessed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Open-label, Single-arm
Number analyzed (Participants) | 16
percentage of participants | 68.8 [46.0 to 91.5]

2. Secondary Outcome: Number of Participants With Grade 3-4 Acute Toxicities
Description: To characterize safety by evaluating Grade 3-4 acute toxicities of adjuvant durvalumab with radiotherapy in intermediate-risk Head and Neck Squamous Cell Carcinoma patients receiving adjuvant durvalumab with radiotherapy. Toxicity was assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE v4.03).
Time Frame: Up to 30 days
Population: Participants started to study the treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label, Single-arm
Number analyzed (Participants) | 16
Participants | 1

3. Secondary Outcome: Chronic Toxicities of Adjuvant Durvalumab With Radiotherapy
Description: To characterize the Grade 3-4 chronic toxicities of adjuvant durvalumab with radiotherapy in intermediate-risk Head and Neck Squamous Cell Carcinoma patients. Toxicity was assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE v4.03).
Time Frame: 12 weeks
Population: The type of Grade 3 Adverse Events observed in 5 subjects were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label, Single-arm
Number analyzed (Participants) | 16
Participants
  Grade 3- Weight loss | 1
  Grade 3- Mucositis oral | 1
  Grade 3- Hypertension | 1
  Grade 3- wrist pain | 1
  Grade 3-Dysphagia | 1
  Grade 3- Lymphedema | 1
  Grade 3- Odynophagia | 1

4. Secondary Outcome: Overall Survial in Patients With Intermediate-risk HNSCC Treated With Adjuvant Durvalumab With Radiotherapy PD-L1 Expression With Disease Free Survival
Description: To estimate median OS in patients with intermediate-risk HNSCC treated with adjuvant durvalumab with radiotherapy.-To correlate PD-L1 expression with disease free survival
Time Frame: 5 years
Reporting Status: Not Posted

5. Secondary Outcome: PD-L1 Expression With Disease Free Survival.
Description: To correlate PD-L1 expression with disease free survival.
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2027-05

ADVERSE EVENTS:
Time Frame: Adverse events were collected from day one of the study drug administration to 30 days after completion of treatment. (Up to 3 years)
Description: National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE v4.03).
Groups:
- Open-label, Single-arm: Durvalumab in combination with intensity-modulated radiotherapy (IMRT) treatments
Arm/Group | Open-label, Single-arm
All-Cause Mortality (participants affected / at risk) | 3/18
Serious Adverse Events (participants affected / at risk) | 1/18
Other Adverse Events (participants affected / at risk) | 17/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label, Single-arm (N=18)
Vascular Disorders - Other, Specify (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label, Single-arm (N=18)
Anemia (Blood and lymphatic system disorders) | 1
Ear And Labyrinth Disorders - Other, Specify (Ear and labyrinth disorders) | 1
Hearing Impaired (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Hyperthyroidism (Endocrine disorders) | 2
Hypothyroidism (Endocrine disorders) | 1
Dry Mouth (Gastrointestinal disorders) | 4
Dysphagia (Gastrointestinal disorders) | 1
Esophageal Stenosis (Gastrointestinal disorders) | 1
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1
Gastrointestinal Disorders - Other, Specify (Gastrointestinal disorders) | 1
Mucositis Oral (Gastrointestinal disorders) | 1
Oral Pain (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 3
Pain (General disorders) | 1
Infections And Infestations - Other, Specify (Infections and infestations) | 1
Alanine Aminotransferase Increased (Investigations) | 1
Aspartate Aminotransferase Increased (Investigations) | 1
Blood Bilirubin Increased (Investigations) | 1
Lipase Increased (Investigations) | 1
Lymphocyte Count Decreased (Investigations) | 7
Serum Amylase Increased (Investigations) | 2
Weight Loss (Investigations) | 3
White Blood Cell Decreased (Investigations) | 2
Hyponatremia (Metabolism and nutrition disorders) | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 1
Fibrosis Deep Connective Tissue (Musculoskeletal and connective tissue disorders) | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 4
Nervous System Disorders - Other, Specify (Nervous system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Laryngeal Edema (Respiratory, thoracic and mediastinal disorders) | 1
Nail Loss (Skin and subcutaneous tissue disorders) | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1
Skin And Subcutaneous Tissue Disorders - Other, Specify (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 2
Lymphedema (Vascular disorders) | 3
Vascular Disorders - Other, Specify (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Subcontractor agrees that the first publication of the Study results will be made by Institution as a multi-site publication. Subcontractor can publish its site-specific results after Institution's publication, 12 months post-study completion, or upon Institution's notice of completion. Subcontractor must provide Institution 30 days for manuscript review and may delay publication for 45 days for institution's patent filing. Institution will register the Study and post results as required by law.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/22/NCT03529422/Prot_SAP_000.pdf